CLINICAL TRIAL: NCT04798235
Title: Phase 1/2, Open-Label Clinical Study to Evaluate the Safety and Efficacy of Intrathecal TSHA-101 Gene Therapy for Treatment of Infantile Onset GM2 Gangliosidosis
Brief Title: First-in-Human Study of TSHA-101 Gene Therapy for Treatment of Infantile Onset GM2 Gangliosidosis
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dr. Anupam Sehgal (Other)
Collaborators: Taysha Gene Therapies, Inc. (Industry); GlycoNet (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Anupam Sehgal, Primary Investigator, Queen's University
Organization: Queen's University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSHA-101-IST-001
Record Dates: First submitted 2021-02-22; First posted 2021-03-15 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Infantile GM2 Gangliosidosis (Disorder)
Keywords: Tay-Sachs disease; Sandhoff disease; GM2 gangliosidosis
MeSH Terms: conditions — Tay-Sachs Disease; Sandhoff Disease; Gangliosidoses, GM2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TSHA-101 (Experimental): Subjects who will receive one-time intrathecal TSHA-101, brain volume based sliding scale for dosage
  Interventions: Biological: TSHA-101

INTERVENTIONS:
Biological: TSHA-101 — AAV9 viral vector containing HEXA and HEXB genes to be administered via Intrathecal injection

SUMMARY:
GM2 gangliosidoses are a group of autosomal recessive neurodegenerative diseases characterized by a deficiency of the Hex A enzyme to catabolize GM2, thereby causing GM2 accumulation within cellular lysosomes.Hex A is composed of 2 subunits, α- and β-, coded by the HEXA and HEXB genes, respectively. The primary purpose of the current study is to assess the safety and tolerability of TSHA101 administered via IT injection.

ELIGIBILITY:
Key Inclusion Criteria:

* male or female with age less than or equal to 15 months
* diagnosis of GM2 gangliosidosis with genetic and enzymatic documentation of infantile disease

Key Exclusion Criteria:

* a second neurodevelopmental disorder independent of the HEXA or HEXB
* inability to tolerate sedation or intrathecal administration
* invasive ventilatory support
* concomitant illness, allergies or known hypersensitivity to the required immunosuppression regimen

Max Age: 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2027-03-12 (Estimated); Study Completion 2027-03-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability: Treatment-emergent Adverse Events (TEAEs) | 1 year
  Incidence, severity, and relatedness of TEAEs
Safety and Tolerability: Number of participants with abnormal Laboratory assessments | 1 year
  Number of participants with Changes from Baseline in laboratory assessments
Safety and Tolerability: Electrocardiogram (ECG) | 1 year
  Changes from Baseline in 12-lead ECG findings in QT interval

SECONDARY OUTCOMES:
Safety and tolerability: Viral shedding analysis | 1 year
  Positive presence of viral DNA from biological fluids (whole blood, urine, saliva, and stool)
Assessment of Immunogenicity: Biomarkers in serum | 1 year
  Summary of neutralizing antibodies (NAbs) titers for adeno-associated virus, serotype 9 (AAV9) and Hex A
Assessment of Immunogenicity: Biomarkers in serum | 1 year
  Summary of total antibodies (TAbs) titers for AAV9 and Hex A
Assessment of Immunogenicity: Biomarkers in peripheral blood mononuclear cells (PBMCs | 5 years
  Summary of PBMCs for enzyme-linked immune absorbent spot (ELISpot) assays for cytokine secretion against AAV9 and Hex A
Overall Survival | treatment to death from any cause, up to 5 years
  Estimated using the Kaplan-Meier method
Hex A Enzyme Activity: Cerebrospinal fluid (CSF) and serum | 1 year
  Change from baseline
Head Control: Number of events for abnormal head control | 1 year
  change from Baseline
Change from Baseline in motor function: Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP-INTEND) | 1 year
  The test consists of 16 items (body parts), where each item is tested for both sides of the body, left and right. The best score is taken for each item (with a maximum score of 4), and the scores are summed over all 16 items with a possible total CHOP-INTEND score of 64.
Change from Baseline in Motor Function: Modified Ashworth Scale | 1 year
  change from Baseline. Increase or decrease of muscle tone will be measured by the Modified Ashworth Scale. Frequency counts and percentages will be presented by score (0, 1, 1+, 2, 3, and 4), muscle, side, and visit for the safety population. Flexion and extension of the knee and elbow will be measured on both sides, along with hip adduction and abduction on both sides of the body.
Clinical Efficacy Assessment: Progression of Hypotonia | 1 year
  Assessed through neurological examinations as present or absent. Baseline to each post-Baseline visit
Clinical Efficacy Assessment: Dysphagia | From onset up to 3 years, if present
  Assessment of the dysphagia events- assessed as present or absent.

CONTACTS AND LOCATIONS:
Overall Officials: Anupam Sehgal, MBBS, Principal Investigator — Queen's University
Locations (1):
- Queen's University/Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ryckman AE, Deschenes NM, Quinville BM, Osmon KJL, Mitchell M, Chen Z, Gray SJ, Walia JS. Intrathecal delivery of a bicistronic AAV9 vector expressing beta-hexosaminidase A corrects Sandhoff disease in a murine model: A dosage study. Mol Ther Methods Clin Dev. 2023 Dec 5;32(1):101168. doi: 10.1016/j.omtm.2023.101168. eCollection 2024 Mar 14. PMID 38205442